CLINICAL TRIAL: NCT03975855
Title: Percutaneous Ultrasound-Guided Biopsy Evaluated for Axillary Lymph Node Sampling Efficacy (PULSE)
Brief Title: Evaluation of NeoNavia® Biopsy System in Axillary Lymph Nodes
Acronym: PULSE
Status: Completed | Type: Observational
Sponsor: NeoDynamics AB (Industry)
Responsible Party: Sponsor
Other Study IDs: NEODOC-2021668610-165
Record Dates: First submitted 2019-05-29; First posted 2019-06-05 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Axillary Lymph Nodes; Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspicious axillary lymph nodes: All patients with histologically confirmed breast cancer or highly suspicious breast lesions presenting with suspicious axillary lymph nodes
  Interventions: Device: NeoNavia® Biopsy System

INTERVENTIONS:
Device: NeoNavia® Biopsy System — Biopsy of axillary lymph node using the NeoNavia Biopsy System. The investigator shall obtain as many/large samples as judged adequate and sufficient for diagnosis.

SUMMARY:
The aim of the study is to document performance characteristics of a biopsy device indicated for use in axillary lymph nodes, to provide basic insights into the complexity of axillary biopsy procedures and generate hypothesis for further larger comparative trials.

This is a Sponsor-initiated prospective, multicenter, registry trial. Patients that present with suspicious axillary lymph nodes at the time of breast cancer diagnosis undergo axillary sampling using the NeoNavia biopsy system. This is in accordance with clinical routine and current clinical guidelines. The system incorporates a new mechanism for controllable and precise needle insertion and a newly developed sampling needle for high yield sampling acquisition. It is approved for use in the breast and axillary lymph nodes.

DETAILED DESCRIPTION:
Determining axillary nodal status at the time of diagnosis is paramount for optimal staging and treatment planning. SLNB is indicated for patients with a clinical and radiological negative axilla. 25%-43% of breast cancer patients are reported to present with radiologically suspicious axillary lymph nodes at the time of diagnosis. In these patients, a pre-operative ultrasound-guided needle sampling of suspicious axillary lymph tissue is indicated.

This can rationalize patient care by identifying those with axillary metastases using merely a minimally-invasive intervention. These patients can be counselled with regards to proceeding directly to definitive axillary surgery in the form of axillary lymph node dissection (ALND) rather than sentinel node biopsy (SLNB), thereby omitting a potentially unnecessary surgical procedure. Patients with a negative axillary status can proceed to SLNB for definitive nodal status determination. Furthermore, in the paradigm of neoadjuvant treatment, confirming a histopathologic involvement of lymph nodes by US-guided needle biopsies enables for decision on neoadjuvant chemotherapy without the need for a surgical procedure.

The main challenge in performing CNB (Core Needle Biopsy) within the axilla is to avoid damaging the major vessels and nerves. Technical, operator and procedural requirements that mitigate risks in CNB sampling of the axilla have been reported in the literature. It is suggested that the operator shall fully acknowledge the detailed anatomy including vessels and nerves in the axilla, have good hand-eye coordination as well as be experienced in US-guided interventions. Proper positioning of the patient is reported to be important. Color Doppler ultrasound shall be used to assess the location of large vessels relative to the intended biopsy track and to avoid sampling a vascular component of the node. Perfect guiding and visualization of the needle tip at all times is reported to be essential. It is suggested that a biopsy device with a controllable needle action is safer to use. Omitting the firing action gives the operator greater control over the final needle tip placement.

Due to the difficulty of the procedure there may be inclusion bias in the reported studies. In one series, patients presenting with nodes adjacent to a vessel or located very deep and difficult to access were not asked to participate in the study and hence not subjected to CNB. In another study FNA (Fine Needle Aspiration) was performed instead of CNB when the lymph nodes were in close proximity to vessels. A recent German survey showed that merely 79% of breast centers (41/52) perform biopsies in the axilla (data on file), and anecdotal evidence suggests that in certain departments only the most experienced physician performs CNB procedures in axillary lymph nodes, risking economic/operational inefficiencies.

For the purpose of documenting the prevalence and composition of cases deemed challenging in this study, an experienced expert panel has compiled a comprehensive list of risk parameters characterizing the anatomic complexity and procedural difficulty of axillary lymph node needle biopsies.

Recently a new biopsy device indicated for the use in breast and axillary lymph nodes (NeoNavia biopsy system, NeoDynamics, Sweden) has become available. It incorporates a pneumatic needle insertion mechanism that is intended to provide better control of needle progression and enable stepwise insertion without noticeable deformation or displacement of surrounding tissue as visualized under ultrasound. Furthermore a new method of tissue acquisition is employed that has pre-clinically shown a higher sampling yield compared to CNB. These characteristics indicate that the device could be well suited for tackling even the most challenging cases of axillary lymph node biopsies. Initial clinical results indicate that in axillary lesions deemed "technically difficult", i.e. where prior US-guided biopsies with CNB or FNA had yielded non-diagnostic histology results, the NeoNavia device performed successfully thereby significantly altering clinical management.

ELIGIBILITY:
Inclusion Criteria:

* cT1-4c (multifocality / multicentricity permitted)
* Female / male patient aged ≥ 18 years
* cN+ based on the following criteria (at least one criteria must be met):

  * lymph node is palpable
  * cortical asymmetry (focal or diffuse cortical thickening of >3mm) under US
  * cortex:hilum ratio >2:1 under US
  * loss of hilum/cortex structure under US
* Written informed consent (ICF)

Exclusion Criteria:

* Suspicious lymph nodes after neoadjuvant therapy
* No confirmed breast cancer and no abnormality in the breast
* Patient uses Marcumar
* Pregnant and lactating women
* Known hypersensitivity reaction against local anesthesia
* Prior chemo or radiation therapy in breast or axilla
* Missing written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from eight university hospitals in Germany
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Rate of successful biopsies (= success rates) | after histopathological analysis af tissue samples, up to 1 week after biopsy
  Lymph node tissue present in biopsy samples as assessed by histopathologist

SECONDARY OUTCOMES:
Rate of patients presenting with risk parameters for an anatomically complex procedure | time of biopsy, 1 day
  Based on a list of parameters established by an expert panel to characterize the anatomic complexity of axillary biopsy procedures
Rate of cases in which it was possible to target the selected lymph node or, if present, the lesion inside the node | time of biopsy, 1 day
Rate of cases in which pulses facilitated control during needle insertion | time of biopsy, 1 day
Sensitivity | post-surgery, up to 200 days
Specificity | post-surgery, up to 200 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Thill, PD Dr., Principal Investigator — Leading Principal Investigator
Locations (7):
- Germany (7):
  - Klinikum Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Universitätsfrauenklinik Tübingen, Tübingen, Baden-Wurttemberg
  - Agaplesion Markus Krankenhaus, Frankfurt am Main, Hesse
  - Universitäts-Frauenklinik, Rostock, Mecklenburg-Vorpommern
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - HJK Erkelenz, Erkelenz, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Essen, North Rhine-Westphalia

REFERENCES:
- [Background] Schassburger KU, Paepke S, Saracco A, Azavedo E, Ekstrom C, Wiksell H. High velocity pulse biopsy device enables controllable and precise needle insertion and high yield tissue acquisition. Phys Med. 2018 Feb;46:25-31. doi: 10.1016/j.ejmp.2017.12.014. Epub 2018 Jan 30. PMID 29519406
- [Background] Gruber I, Hahn M, Fehm T, Hann von Weyhern C, Stabler A, Winckelmann A, Wallwiener D, Kuhn T. Relevance and methods of interventional breast sonography in preoperative axillary lymph node staging. Ultraschall Med. 2012 Aug;33(4):337-43. doi: 10.1055/s-0031-1273317. Epub 2011 May 26. PMID 21618166
- [Background] Nakamura R, Yamamoto N, Miyaki T, Itami M, Shina N, Ohtsuka M. Impact of sentinel lymph node biopsy by ultrasound-guided core needle biopsy for patients with suspicious node positive breast cancer. Breast Cancer. 2018 Jan;25(1):86-93. doi: 10.1007/s12282-017-0795-7. Epub 2017 Jul 22. PMID 28735457
- [Background] Garcia-Ortega MJ, Benito MA, Vahamonde EF, Torres PR, Velasco AB, Paredes MM. Pretreatment axillary ultrasonography and core biopsy in patients with suspected breast cancer: diagnostic accuracy and impact on management. Eur J Radiol. 2011 Jul;79(1):64-72. doi: 10.1016/j.ejrad.2009.12.011. Epub 2010 Jan 4. PMID 20047809
- [Background] Abe H, Schmidt RA, Kulkarni K, Sennett CA, Mueller JS, Newstead GM. Axillary lymph nodes suspicious for breast cancer metastasis: sampling with US-guided 14-gauge core-needle biopsy--clinical experience in 100 patients. Radiology. 2009 Jan;250(1):41-9. doi: 10.1148/radiol.2493071483. Epub 2008 Oct 27. PMID 18955508
- [Background] Kim KH, Son EJ, Kim EK, Ko KH, Kang H, Oh KK. The safety and efficiency of the ultrasound-guided large needle core biopsy of axilla lymph nodes. Yonsei Med J. 2008 Apr 30;49(2):249-54. doi: 10.3349/ymj.2008.49.2.249. PMID 18452262
- [Background] Ganott MA, Zuley ML, Abrams GS, Lu AH, Kelly AE, Sumkin JH, Chivukula M, Carter G, Austin RM, Bandos AI. Ultrasound Guided Core Biopsy versus Fine Needle Aspiration for Evaluation of Axillary Lymphadenopathy in Patients with Breast Cancer. ISRN Oncol. 2014 Feb 4;2014:703160. doi: 10.1155/2014/703160. eCollection 2014. PMID 24649373
- [Background] Damera A, Evans AJ, Cornford EJ, Wilson AR, Burrell HC, James JJ, Pinder SE, Ellis IO, Lee AH, Macmillan RD. Diagnosis of axillary nodal metastases by ultrasound-guided core biopsy in primary operable breast cancer. Br J Cancer. 2003 Oct 6;89(7):1310-3. doi: 10.1038/sj.bjc.6601290. PMID 14520465